CLINICAL TRIAL: NCT04306406
Title: Molecular Mechanisms Underlying the Protective Effects of Whole Red Raspberries Against Insulin Resistance and Inflammation in Type 2 Diabetes
Brief Title: Molecular Mechanisms of Raspberries Effect on Insulin Resistance and Inflammation
Acronym: RASPBERRY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: National Processed Raspberry Council (Unknown); Louisiana State University and A&M College (Other)
Responsible Party: Principal Investigator, Frank Greenway, Professor; Chief Medical Officer, Pennington Biomedical Research Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2015-0004
Record Dates: First submitted 2019-07-30; First posted 2020-03-12 (Actual); Last update posted 2020-03-12 (Actual); Status verified 2020-03

CONDITIONS: Inflammation; Insulin Resistance
MeSH Terms: conditions — Inflammation; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Raspberry Smoothies (Other): Single serving smoothies drink made with red raspberries to be consumed daily for two weeks
  Interventions: Other: Raspberries

INTERVENTIONS:
Other: Raspberries — Red raspberry smoothies drink

SUMMARY:
Red raspberries (Rubus idaeus) are a good source of health enhancing hydrolyzable and condensed tannins, flavonoids, anthocyanins, phenolic acids, rheosmin, potassium, carotenoids, vitamin C, and vitamin K1. Compared to other berries commonly consumed in the US, the health benefits of red raspberries to improve pre-diabetes mellitus (PDM) and type 2 diabetes have never been explored. The clinical study proposed in this project seeks to investigate the protective effect of whole red raspberries against insulin resistance, oxidative stress, and inflammation in PDM and type 2 diabetic patients. The in vitro study proposed in the project will assist in identifying the molecular mechanisms by which whole red raspberry protect islet cells against oxidative stress, insulin resistance and loss of cell function.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes

Exclusion Criteria:

* hypoglycemic agents
* Pregnant or nursing a child
* chronic medication that does not have a stable dose for greater than one month
* anti-inflammatory medication
* inflammatory disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2015-01-07 (Actual); Primary Completion 2017-01-13 (Actual); Study Completion 2017-01-13 (Actual)

PRIMARY OUTCOMES:
Homeostatic Model Assessment for Insulin Resistance (HOMA-IR) | 2 weeks
  Ratio of fasting insulin and glucose
A high-sensitivity C-reactive protein (hs-CRP) measured in milligrams per liter | 2 weeks
  Measure of systemic inflammation

SECONDARY OUTCOMES:
3,4-Dihydroxyphenylacetic acid (DOPAC) measured in nanograms per milliliter | 2 weeks
  Measure of systemic inflammation

CONTACTS AND LOCATIONS:
Overall Officials: Frank L Greenway, MD, Principal Investigator — Pennington Biomedical Research Center

IPD SHARING:
Plan to Share IPD: Yes
Excel spreadsheets containing clinical trial data can be made available to other researchers after publication of research results.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will become available after publication of research results.
Access Criteria: Academic researcher